CLINICAL TRIAL: NCT02664584
Title: The Trinity, Ulster and Department of Agriculture Cohort Study
Acronym: TUDA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Ulster (Other)
Collaborators: University of Dublin, Trinity College (Other); University College Cork (Other); University College Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: 08NIR03/113
Record Dates: First submitted 2016-01-14; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Disease; Osteoporosis; Alzheimer's Disease; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Osteoporosis; Alzheimer Disease; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples Buccal swabs Buffy coats
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cross-sectional cohort: Cohort who took part in the cross-sectional study (n=5186)
- Cross-sectional cohort + follow-up: Cohort who took part in both the cross-sectional and follow-up study (planned n=500 (on-going))

SUMMARY:
Background:

Cardiovascular disease (CVD), osteoporosis and dementia are chronic diseases of ageing that impact adversely on the lives of those affected and have major health, social and economic consequences. A number of factors are considered to be implicated in these diseases, ranging from the more established factors to those that are less well recognised. Lifestyle factors such as diet, body weight, smoking, physical activity and years of education are acknowledged as risk factors for the development of these chronic diseases of aging. Emerging research suggests that elevated homocysteine and/or sub-optimal status of the metabolically related B-vitamins (folate, vitamin B12, B6 and riboflavin) may be associated with a higher risk of age-related disease. The interplay between relevant genetic and nutrient factors (gene-nutrient interactions) is considered to be highly relevant in the development (and prevention) of chronic diseases of ageing, however this relatively new area of research is as yet poorly understood. The collection of clinical, lifestyle, nutritional and genetic data on large numbers of patients would permit the investigation of those nutrients which interact with specific genes to increase the likelihood of a person developing chronic diseases of ageing.

Aim:

The aim of the TUDA study is to collect detailed clinical, lifestyle, dietary, genetic and biochemical data to investigate gene-nutrient interactions (particularly from the perspective of the B-vitamins and vitamin D/calcium) in the development of CVD, osteoporosis and dementia by studying older adults exhibiting the early stages of these common diseases, namely hypertension, low bone mineral density, and early memory loss, respectively.

Secondary aim (follow up TUDA investigation):

The aim of this longitudinal investigation is to re-assess clinical, nutritional, genetic and biochemical factors in relation to the progression of disease outcomes in TUDA study participants, in subsequent years after initial investigation.

Study design:

A total of 6000 non-institutionalised older Irish people aged over 60 years with early predictors of either dementia, stroke and osteoporosis (namely early memory loss, high blood pressure and low bone mineral density, respectively) recruited from three centres (St James's Hospital Dublin, Ulster University Coleraine and The Clinical Translational Research and Innovation Centre (C-TRIC), Londonderry) across Ireland. Non-fasting blood samples were collected from all subjects and routine blood biochemistry profiles and biomarkers of relevance to B vitamin and vitamin D status were measured. Supplement use was recorded and a targeted food frequency questionnaire was used to record dietary intakes of specific vitamins of interest (folate, B12, B6, riboflavin and D) from major food sources, particularly fortified foods. Physiological function tests including blood pressure, bone health (DXA scans) and cognitive function tests and anthropometric measures were also taken.

ELIGIBILITY:
Inclusion Criteria:

* >60 years of age

Exclusion Criteria:

* <60 years of age
* Born outside the island of Ireland
* Severe dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 and above
Sampling Method: Non-Probability Sample
Enrollment: 5186 (Actual)
Dates: Start 2008-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 10 years
Bone health (DXA) | 10 years
  Dual energy x ray absorptiometry (DXA) scan
Cognitive function 1 (MMSE) | 10 years
  Mini-Mental State Examination (MMSE)
Cognitive function 2 (FAB) | 10 years
  Frontal Assessment Battery (FAB)
Cognitive function 3 (RBANS) | 10 years
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Anxiety (HADS) | 10 years
  Hospital Anxiety and Depression Scale (HADS)
Depression (CES-D) | 10 years
  Center for Epidemiologic Studies Depression Scale (CES-D)

SECONDARY OUTCOMES:
Weight | 10 years
Routine biochemical markers | 10 years
  Measured in blood
Vitamin biomarkers | 10 years
  Measured in blood
Single nucleotide polymorphisms | 10 years
  Measured in DNA sample
Measures of mobility (TUG) | 10 years
  Timed Up and Go (TUG)
Measures of muscle strength | 10 years
  Hand grip strength (dynamometer)
Bone turnover markers | 10 years
  Measured in blood

CONTACTS AND LOCATIONS:
Locations (3):
- St James's Hospital, Dublin, Dublin8, Ireland
- United Kingdom (2):
  - Human Intervention Studies Unit, Ulster University, Coleraine, Londonderry
  - Clinical Translational Research and Innovation Centre (C-TRIC), Altnagelvin Hospital, Londonderry, Londonderry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon S, Hoey L, McNulty H, Keenan J, Pangilinan F, Brody LC, Ward M, Strain JJ, McAnena L, McCann A, Molloy AM, Cunningham C, McCarroll K, Hughes CF. Associations of one-carbon metabolism, related B-vitamins and ApoE genotype with cognitive function in older adults: identification of a novel gene-nutrient interaction. BMC Med. 2025 Jul 28;23(1):440. doi: 10.1186/s12916-025-04276-8. PMID 40717068
- [Derived] Jarrett H, McNulty H, Hughes CF, Pentieva K, Strain JJ, McCann A, McAnena L, Cunningham C, Molloy AM, Flynn A, Hopkins SM, Horigan G, O'Connor C, Walton J, McNulty BA, Gibney MJ, Lamers Y, Ward M. Vitamin B-6 and riboflavin, their metabolic interaction, and relationship with MTHFR genotype in adults aged 18-102 years. Am J Clin Nutr. 2022 Dec 19;116(6):1767-1778. doi: 10.1093/ajcn/nqac240. PMID 36264281